CLINICAL TRIAL: NCT00184249
Title: A Prospective Multi Centre Trial on Bipolar Radiofrequency Ablation of Atrial Fibrillation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Collaborators did not enter patients into the study
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Oslo University Hospital (Other); Haukeland Sykehus HF (Unknown); Ullevaal University Hospital (Other); Regionssykehuset i Tromsø HF (Unknown); Feiringklinikken (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120905
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Atrial Fibrillation
Keywords: Catheter ablation; Heart/surgery; Cardial surgical procedures
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bipolar radiofrequency ablation (Experimental)
  Interventions: Procedure: Bipolar radiofrequency ablation

INTERVENTIONS:
Procedure: Bipolar radiofrequency ablation — Ablation using CE marked bipolar ablation devices
  Other Names: Cardioblade; Atricure

SUMMARY:
The study is a prospective multi-centre study to investigate the effect of a new bipolar ablation strategy of the left atrium in patients with paroxysmal or permanent atrial fibrillation over time.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common persistent arrhythmia, prevalent in about 6% of the population over 65 years of age. AF reduces the quality of life and increases mortality. AF is particularly common in combination with mitral valve disease, but is also detected in about 5% of patients with aortic valve and coronary artery disease. Surgical treatment of AF with the Cox-maze III operation was developed by J. Cox during the 80ies. The aim of the operation is to block spread of irregular electrical activity by creating lines of isolation in the atrial musculature. The operation achieves sinus rhythm in over 90% in selected patients. Nevertheless the method was only used in few heart surgical centres, because it is complex and time consuming.In recent years alternative energy sources have been developed to create isolating lines without cutting the tissue and thus making ablation treatment easier. Bipolar radiofrequency ablation is special because the energy is delivered feedback controlled until transmurality is achieved. This is a prerequisite for a good result and makes using the equipment safer.

Since the development of the Cox-maze procedure, our knowledge of atrial fibrillation and its treatment has increased considerably. There is a consensus that the posterior part of the left atrium and in particular the pulmonary veins are an important target for treatment. Surgical ablation with alternative energy sources is a new method under continued development and evaluation.

The optimal ablation treatment is unknown. A balance between invasiveness and achieving sinus rhythm in as many as possible has to be found. Creating numerous ablation lines in both atria is time consuming and leads probably to an increased need for permanent pacemaker implantation and reduced contractility of the atrial tissue. On the other hand can a simple bipolar ablation of pulmonary veins performed easily, but this is probably an insufficient treatment for most patients. In the protocol a new method using solely bipolar ablation for creation of several ablation lines in the left atrium is described.

The study is a prospective multi-centre study to investigate the effect of a new bipolar ablation strategy of the left atrium in patients with paroxysmal or permanent AF over time.

ELIGIBILITY:
Inclusion Criteria:

* referred for elective heart surgery with extracorporeal circulation
* suffers from AF for more than 6 months but less than 7 years
* aged between 18 and 80 years
* ejection fraction above 30 %

Exclusion Criteria:

* Reoperations
* NYHA class IV
* Ischemic mitral incompetence
* Creatinine > 140
* Transmural myocardial infarction < 4 weeks
* Endocarditis
* Serious peripheral vascular disease
* Pregnancy or breast-feeding
* Drug addiction
* Size of left atrium > 60 mm in preoperative echo-doppler investigation.
* Disease or other condition when the patient is unable to understand the objectives and the scope of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-06; Primary Completion 2010-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Number of patients in sinus rhythm after 3, 6, and 12 months | 3, 6,
Number of patients with atrial function at echo-doppler after 6 and 12 months | 3,6, 12 months
Number of patients on anticoagulants after 6 and 12 months | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Wahba, Prof, Study Director — Norwegian University of Science and Technology